CLINICAL TRIAL: NCT01730976
Title: Asthma in the Elderly: The Role of Vitamin D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C. (Other)
Responsible Party: Principal Investigator, Michele Columbo, M.D., Principal Investigator, Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F/N-R13-3217B; SSRF2012-01 (Other Grant/Funding Number: SSRF2012-01)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Asthma in the Elderly
Keywords: asthma, elderly, vitamin D
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D 2,000 I.U. daily (Experimental): Study subjects will take 2,000 I.U. vitamin D daily for three months
  Interventions: Dietary Supplement: Vitamin D 2,000 I.U.

INTERVENTIONS:
Dietary Supplement: Vitamin D 2,000 I.U.
  Other Names: Vitamin Shoppe

SUMMARY:
We will study whether taking vitamin D improves asthma control and spirometric values in elderly asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Asthma, age of 65 years old or older

Exclusion Criteria:

* Current smokers, subjects who smoked more than 10 pack/year, subjects taking digoxin, subjects with liver disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Asthma Control Test (ACT) score | Three months

SECONDARY OUTCOMES:
Improvement in pulmonary function tests values (FEV1%, etc.) | Three months

OTHER OUTCOMES:
Serum vitamin D and calcium levels | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Columbo, M.D., Principal Investigator — Rohr and Columbo Associates
Locations (1):
- Rohr and Columbo Asthma, Allergy and Immunology Specialists, Bryn Mawr, Pennsylvania, United States

REFERENCES:
- [Derived] Columbo M, Panettieri RA Jr, Rohr AS. Asthma in the elderly: a study of the role of vitamin D. Allergy Asthma Clin Immunol. 2014 Sep 5;10(1):48. doi: 10.1186/1710-1492-10-48. eCollection 2014. PMID 25221606